CLINICAL TRIAL: NCT03627117
Title: Randomized Placebo Controlled Cross-over Study Investigating the Influence of CBD on Episodic Memory in Healthy Subjects
Brief Title: Influence of CBD on Episodic Memory in Healthy Subjects
Acronym: CoIL-Basel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dominique de Quervain, MD (Other)
Responsible Party: Sponsor-Investigator, Prof. Dominique de Quervain, MD, Prof. Dr. med., University of Basel
Organization: University of Basel (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2018-01125
Record Dates: First submitted 2018-07-11; First posted 2018-08-13 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Healthy
MeSH Terms: interventions — calcium D-pantothenate, L-cysteine drug combination

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum/Placebo (Experimental): This group will start with CBD and after washout will receive placebo.
  Interventions: Drug: Verum; Drug: Placebo
- Placebo/Verum (Experimental): This group will start with placebo and will receive CBD after washout.
  Interventions: Drug: Verum; Drug: Placebo

INTERVENTIONS:
Drug: Verum — Single vape of 0.25mL of CBD e-Liquid containing: 5% CBD (low-temperature extracted Cannabidiol from Cannabis sativa L., purity 99%), Glycerine (vegetable), Propylene glycol, water
  Other Names: Cannabidinol (CBD) e-Liquid
Drug: Placebo — Single vape of 0.25ml e-liquid La Baronne Jaune, BORDO2.
  Other Names: e-Liquid

SUMMARY:
Placebo controlled, randomized, double blind, cross-over design.

Single vape of 0.25ml 5% CBD e-liquid (12.5mg CBD) and single vape of 0.25ml e-liquid, tastes like lemon and madeleine. 15min vape time each.

A total of 34 participants, equal number of male and female. There will be replacement of Drop-Outs until data from 34 participants are completed.

The primary endpoint will be performance in a verbal memory task. The secondary endpoint will be performance in a working memory test.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Normotensive (BP between 90/60mmHg and 140/90mmHg)
* BMI between 18 and 30 kg/m2
* Male or female
* Aged between 18 and 30 years
* Native or fluent German-speaking
* Able and willing to give written informed consent as documented by signature and comply with the requirements of the study protocol
* Willing to donate urine sample to control for pre-Visit CBD/THC consume

Exclusion Criteria:

* Acute or chronic psychiatric disorder including drug or alcohol abuse
* Women who are pregnant or breast feeding
* Intention to become pregnant during the course of the study
* Smoking (> 5 cigarettes per day)
* Participation in one of our previous studies using the same verbal test in the past 2 years
* Participation in a study with CBD / THC within the 30 days preceding and during the present study
* Known hypersensitivity or allergy to propylene glycol
* Intake of CBD / THC within the 7 days preceding and during the present study in any application form
* Long-term systemic medication or topical steroids to treat an underlying disease within last 3 months
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2018-12-08 (Actual); Study Completion 2018-12-08 (Actual)

PRIMARY OUTCOMES:
Verbal memory task | Timepoint 21 minutes after first medication.
  Three series of five semantically unrelated nouns will be presented. Total score is calculated by summing the number of correctly recalled words. Higher scores represent a better outcome. Score Minimum 0 and score maximum 15.

SECONDARY OUTCOMES:
Working memory | Timepoint 15 minutes after medication.
  Working memory will be assessed by means of a letter 0-back and 2-back task (Papassotiropoulos et al., 2011). The 0-back condition serves as a low-load control condition, measuring general attention and does not require the manipulation of information within working memory. In the 2-back condition, participants have to compare the currently presented letter with the one presented 2 steps before and have to indicate whether they are identical or not. The 2-back condition requires online monitoring, updating and manipulation of remembered information and therefore is assumed to involve key processes of working memory. Accuracy and reaction time will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Janine Hotz, Study Chair — Universität Basel, Birmannsgasse 8, CH-4055 Basel
Locations (1):
- University of Basel, Division of Cognitive Neuroscience, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-11): https://cdn.clinicaltrials.gov/large-docs/17/NCT03627117/Prot_SAP_000.pdf